CLINICAL TRIAL: NCT04989283
Title: NASSIST (Neoadjuvant Chemoradiation +/- Immunotherapy Before Surgery for Superior Sulcus Tumors): A Randomized Phase II Trial of Trimodality +/- Atezolizumab in Resectable Superior Sulcus Non-Small Cell Lung Cancer
Brief Title: Testing the Addition of an Immunotherapy Drug, Atezolizumab, to the Usual Chemotherapy Treatment During Radiation Therapy for Superior Sulcus Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to no accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-08318; NCI-2021-08318 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1934 (Other: SWOG); S1934 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2021-08-03; First posted 2021-08-04 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IIB Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Superior Sulcus Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Biopsy; Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Congresses as Topic; Radiation; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (atezolizumab, chemotherapy, RT, surgery) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1. Patients also receive one of the chemotherapy combinations below depending on their previous therapy and disease. Between the first day of chemotherapy and the first day of cycle 2 of chemotherapy, patients undergo external beam radiation therapy 5 days per week. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning 21 and 90 days after treatment, patients undergo surgery. Within 42 days after completion of surgery, patients then receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients may undergo a PET scan, CT scan, and MRI on study. Patients also undergo tumor biopsies and blood sample collection throughout the trial.
  Interventions: Biological: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery
- Arm II (chemotherapy, RT, surgery) (Active Comparator): Patients receive one of the chemotherapy combinations below depending on their previous therapy and disease. Between the first day of chemotherapy and the first day of cycle 2 of chemotherapy, patients also undergo external beam radiation therapy 5 days per week. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning 21 and 90 days after treatment, patients undergo surgery. Patients may undergo a PET scan, CT scan, and MRI on study. Patients also undergo tumor biopsies and blood sample collection throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
  Arms: Arm I (atezolizumab, chemotherapy, RT, surgery)
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP16
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial tests the effect of atezolizumab given with usual chemotherapy during radiation therapy in treating patients with superior sulcus non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as cisplatin, carboplatin, etoposide, paclitaxel and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Giving atezolizumab with usual chemotherapy and radiation therapy may lower the chance of the tumor from growing or spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the pathologic complete response (pCR) by local review between participants randomized to conventional trimodality therapy, with or without atezolizumab.

SECONDARY OBJECTIVES:

I. To compare event-free survival (EFS) between the arms. II. To compare overall survival (OS) between the arms. III. To compare surgical resection rate and complete resection (R0) rate between the arms.

IV. To evaluate progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 among participants who do not undergo surgical resection, by treatment arm.

V. To compare the frequency and severity of toxicities between the arms.

ADDITIONAL OBJECTIVES:

I. To bank blood and tissue for future research. II. To evaluate the association between major pathologic response (MPR), as defined by the International Association for the Study of Lung Cancer (IASLC), and survival outcomes (OS, PFS).

III. To evaluate the association between pCR by centralized review and survival outcomes (OS, PFS).

IV. Evaluate the changes in fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) metrics (e.g., standardized uptake value [SUV] maximum [max], SUVpeak, SUVmax tumor-to-liver, SUVpeak tumor-to-liver, metabolic tumor volume, total lesion glycolysis, etc.) in participants randomized to receive trimodality therapy alone or in combination with atezolizumab and to evaluate the association with pCR.

V. Evaluate the extent to which the changes in diffusion weighted imaging (DWI)-magnetic resonance imagining (MRI) metrics (e.g., mean apparent diffusion coefficient or apparent diffusion coefficient [ADC] for the primary tumor, etc.) are associated with pCR in participants randomized to receive trimodality therapy alone or in combination with atezolizumab.

VI. Evaluate the extent to which changes in computed tomography (CT) tumor volume, unidimensional lesion changes per RECIST 1.1 and bidimensional lesion changes per World Health Organization (WHO) criteria are associated with pCR in participants randomized to receive trimodality therapy alone or in combination with atezolizumab.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1. Patients also receive one of the chemotherapy combinations below depending on their previous therapy and disease. Between the first day of chemotherapy and the first day of cycle 2 of chemotherapy, patients undergo external beam radiation therapy 5 days per week. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning 21 and 90 days after treatment, patients undergo surgery. Within 42 days after completion of surgery, patients then receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive one of the chemotherapy combinations below depending on their previous therapy and disease. Between the first day of chemotherapy and the first day of cycle 2 of chemotherapy, patients also undergo external beam radiation therapy 5 days per week. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning 21 and 90 days after treatment, patients undergo surgery.

Patients receive one of the chemotherapy combinations:

1. Cisplatin IV over 2 hours on day 1 and etoposide IV over 30-60 minutes on days 1-3.
2. Carboplatin IV over 60 minutes on day 1 and etoposide IV over 30-60 minutes on days 1-3.
3. Paclitaxel IV over 3 hours and carboplatin IV over 60 minutes on day 1.

   Patients with non-squamous NSCLC may receive one of the following combinations:
4. Pemetrexed IV over 10 minutes and carboplatin IV over 60 minutes on day 1.
5. Pemetrexed IV over 10 minutes and cisplatin IV over 2 hours on day 1.

Patients may undergo a PET scan, CT scan, and MRI on study. Patients also undergo tumor biopsies and blood sample collection throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 RANDOMIZATION: Participants must have histologically confirmed cT3/T4, N0/1, M0 non-small cell lung cancer (NSCLC) of the superior sulcus arising in the apex of the lung, involving apical chest wall structures (parietal pleura and beyond) above the level of the second rib
* STEP 1 RANDOMIZATION: Participants must have eligibility affirmed by a thoracic surgeon, medical oncologist and radiation oncologist. Participant must be a candidate for surgical resection and chemoradiation therapy. The site treating investigator must sign off to indicate that eligibility has been affirmed by each specialist
* STEP 1 RANDOMIZATION: Participants may have measurable or non-measurable disease. Measurable disease must be assessed within 28 days prior to Step 1 Randomization. Non-measurable disease must be assessed within 42 days prior to Step 1 Randomization. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form
* STEP 1 RANDOMIZATION: Participants must have an MRI or CT scan of the brain (with contrast highly recommend) within 42 days prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants must have a CT (chest with contrast highly recommended), contrast MRI (thoracic inlet), and FDG-PET/CT performed within 28 days prior to Step 1 Randomization

  * Note: DWI (Diffusion weighting imaging) is highly recommended on the MRI
* STEP 1 RANDOMIZATION: Participants may participate in concomitant non-therapeutic trials (e.g., palliative care assessment or quality of life studies)
* STEP 1 RANDOMIZATION: History and physical exam must be obtained within 28 days of Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants must have Zubrod performance status of 0-1 documented within 28 days prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants must be >= 18 years old
* STEP 1 RANDOMIZATION: Leukocytes >= 3,000/uL (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Absolute neutrophil count >= 1,500/uL (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Platelets >= 100,000/uL (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Participants with known Gilbert disease: total bilirubin =< 3 x (ULN) (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional ULN (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Hemoglobin >= 9 g/dL (within 28 days prior to Step 1 Randomization)
* STEP 1 RANDOMIZATION: Participants must not have higher than grade 2 hypercalcemia prior to Step I Randomization
* STEP 1 RANDOMIZATION: Participants must have a serum creatinine =< the institutional upper limit of normal (IULN) OR measured OR calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants with known human immunodeficiency virus (HIV)-infection must be receiving anti-retroviral therapy and have undetectable viral load test within 6 months prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load within in 28 days prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants of reproductive potential must have a negative serum pregnancy test within 14 days prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants must be offered the opportunity to participate in specimen banking
* STEP 1 RANDOMIZATION: Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
* STEP 2 SURGERY: Participants must have a CT scan of the chest with contrast, FDG-PET/CT scan and MRI scan of the thoracic inlet (with intravenous contrast and DWI highly recommended) within 28 days prior to Step 2 Registration
* STEP 2 SURGERY: Participants must be evaluated for appropriateness of surgery by a thoracic surgeon within 6 weeks after completion of neoadjuvant therapy prior to Step 2 Registration
* STEP 2 SURGERY: Participant's surgery must occur between 21 and 90 days following the end of participant's final cycle of chemotherapy +/- atezolizumab
* STEP 2 SURGERY: Participants must have received at least two cycles of all assigned protocol drugs during neoadjuvant protocol treatment and must have received at least 45 GY RT of the planned 61.2 GY RT during neoadjuvant protocol treatment
* STEP 2 SURGERY: Participants must have a Zubrod Performance Status of 0-1 documented within 28 days prior to Step 2 Registration
* STEP 2 SURGERY: Participants must have postoperative predicted forced expiratory volume in 1 second (FEV1) > 35% and postoperative predicted diffusion capacity of the lung for carbon monoxide (DLCO) > 35%. Pulmonary function tests to ascertain these values must be obtained within 28 days prior to Step 2 Registration
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Participants must have received surgical resection of the lung cancer and side effects must have recovered to =< grade 2 within 42 days after surgery and prior to Step 3 Registration
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Participants must have a Zubrod Performance Status of 0-1 documented within 28 days prior to Step 3 Registration
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Leukocytes >= 3,000/uL (within 28 days prior to Step 3 Registration)
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Absolute neutrophil count >= 1,000/uL (within 28 days prior to Step 3 Registration)
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Platelets >= 100,000/uL (within 28 days prior to Step 3 Registration)
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Hemoglobin >= 9 g/dL (within 28 days prior to Step 3 Registration)
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Total bilirubin =< institutional upper limit of normal (ULN) (within 28 days prior to Step 3 Registration)
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): AST and ALT =< 3 x institutional ULN (within 28 days prior to Step 3 Registration)
* STEP 3 MAINTENANCE THERAPY (ARM 1 ONLY): Participants must have adequate kidney function defined as creatinine =< 1.5 x ULN documented within 28 days prior to Step 3 Registration

Exclusion Criteria:

* STEP 1 RANDOMIZATION: Participants must not have had prior therapy for this cancer including surgery, chemotherapy, immunotherapy, targeted therapy agent, and/or radiation therapy
* STEP 1 RANDOMIZATION: Participants must not have undergone prior radiation to overlapping regions of planned protocol radiation therapy (RT) treatment area
* STEP 1 RANDOMIZATION: Participants must not have had prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* STEP 1 RANDOMIZATION: Participants must not have had prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks prior to Step 1 Randomization
* STEP 1 RANDOMIZATION: Participants must not have a known allergy or hypersensitivity to any component of the carboplatin, pemetrexed, cisplatin, etoposide and paclitaxel formulation
* STEP 1 RANDOMIZATION: Participants must not have any grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., participants with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 3 months, or serious uncontrolled cardiac arrhythmia
* STEP 1 RANDOMIZATION: Participants must not have known active tuberculosis (TB)
* STEP 1 RANDOMIZATION: Participants must not have uncontrolled non-malignant pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (more than once a month). Note: Participants with indwelling catheters (e.g., PleurX [registered trademark]) are allowed
* STEP 1 RANDOMIZATION: Patients must not have undergone prior allogeneic stem cell transplantation or prior solid organ transplantation
* STEP 1 RANDOMIZATION: Participants must NOT have a history of severe allergic, anaphylactic, or other known hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* STEP 1 RANDOMIZATION: Participants must NOT have a known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* STEP 1 RANDOMIZATION: Participants must not have severe or active infections within 28 days prior to Step 1 Randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* STEP 1 RANDOMIZATION: Participants must not have active autoimmune disease requiring therapy within the past 6 months. Participants must not have active autoimmune disease that has required systemic treatment within the past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Autoimmune diseases include, but are not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. This protocol includes an immunotherapy agent which can precipitate known autoimmune diseases
* STEP 1 RANDOMIZATION: Participants must not have history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (e.g., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis. This protocol includes an immunotherapy agent which can precipitate known pneumonitis
* STEP 1 RANDOMIZATION: Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* STEP 1 RANDOMIZATION: Participants must not have received a live attenuated vaccination within 28 days prior to Step 1 Randomization. All coronavirus disease 2019 (COVID-19) vaccines that have received Food and Drug Administration (FDA) approval or FDA emergency use authorization are acceptable
* STEP 1 RANDOMIZATION: Participants must not have had a major surgery within 14 days prior to Step 1 Randomization. Participants must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* STEP 1 RANDOMIZATION: Participants must not be pregnant or nursing due to carcinogenic and teratogenic effects of treatment. Women/men of reproductive potential must have agreed to use an effective contraceptive method while on study treatment and for 5 months after the last dose. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined, he/she is responsible for beginning contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-09 (Estimated); Primary Completion 2031-05-10 (Estimated); Study Completion 2031-05-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) by local review | Up to 6 years

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 6 years
  Defined as From date of Step1 Randomization to date of first documentation of progression that renders participant unable to receive planned protocol surgery, off protocol therapy for any reason without subsequent protocol surgery, relapse after surgery, symptomatic deterioration or death due to any reason, whichever comes first. The primary analysis of EFS will be done using a 1-sided 15% level log-rank test. Will be estimated using the method of Kaplan-Meier. 95% confidence intervals for the medians will be constructed using the method of Brookmeyer-Crowley. Fine-Gray method will be used for a competing risk analysis.
Overall survival (OS) | From date of Step 1 Randomization to date of death due to any cause, assessed up to 6 years
  Will be estimated using the method of Kaplan-Meier. 95% confidence intervals for the medians will be constructed using the method of Brookmeyer-Crowley.
Surgical resection rate | Up to 6 years
Complete resection (R0) rate | Up to 6 years
Progression-free survival (PFS) | From date of Step 1 Randomization to date of first documentation of progression or symptomatic deterioration, or death due to any cause, whichever comes first, assessed up to 6 years
  Will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be estimated using the method of Kaplan-Meier. 95% confidence intervals for the medians will be constructed using the method of Brookmeyer-Crowley.
Incidence of adverse events | Up to 6 years
  Will compare the frequency and severity of toxicities between the arms.

OTHER OUTCOMES:
Bank blood and tissue for future research | Up to 6 years
Major pathologic response | Up to 6 years
  Defined by the International Association for the Study of Lung Cancer, will be associated with and survival outcomes (OS, PFS).
pCR by centralized review | Up to 6 years
  Will be associated with survival outcomes (OS, PFS).
Changes in fludeoxyglucose F-18-positron emission tomography metrics | Baseline up to 6 years
Changes in diffusion weighted imaging (DWI)-magnetic resonance imagining (MRI) metrics | Baseline up to 6 years
  Changes in DWI-MRI metrics will be associated with pCR between arms.
Changes in computed tomography tumor volume | Baseline up to 6 years
  Will assess unidimensional lesion changes per RECIST 1.1 and bidimensional lesion changes per World Health Organization (WHO) criteria. Will be associated with pCR in participants randomized to receive trimodality therapy alone or in combination with atezolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond U Osarogiagbon, Principal Investigator — SWOG Cancer Research Network
Locations (46):
- United States (46):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm